CLINICAL TRIAL: NCT04418843
Title: Cold EMR Vs Standard EMR for the Treatment of Large Nonpedunculated Homogeneous Colorectal Lesions.Randomized and Multicentric Clinical Trial
Brief Title: Cold EMR Vs Standard EMR for the Treatment of Large Nonpedunculated Homogeneous Colorectal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oscar Nogales (Other)
Collaborators: Spanish Society of Digestive Endoscopy (Other)
Responsible Party: Sponsor-Investigator, Oscar Nogales, Principal Investigator, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMEFRÍA.2019
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Adenoma Colon; Serrated Polyp; Serrated Adenoma; Colorectal Neoplasms
Keywords: endoscopic mucosal resection; cold snare endoscopic mucosal resection; standard endoscopic mucosal resection; large nonpedunculated homogeneous colorectal lesions; adenoma colon; serrated polyp; serrated adenoma; conventional endoscopic mucosal resection; laterally spreading adenomas.
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective randomized study (1:1), multicenter, non-blind of consecutive non-pedunculated lesions of serrated and adenomatous histology, homogeneous, with a size greater than or equal to 20 mm (no upper limit in size). Performing cold-EMR vs standard EMR. A non-inferiority study of cold-EMR versus standard EMR.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Endoscopic Mucosal Resection (Experimental): Standard Endoscopic Mucosal Resection, if necessary, multi-piece to resect large nonpedunculated homogeneous colorectal lesions (>20 mm)
  Interventions: Procedure: Standard Endoscopic Mucosal Resection
- Cold Snare Endoscopic Mucosal Resection (Experimental): Cold Snare Endoscopic Mucosal Resection, if necessary, multi-piece to resect large nonpedunculated homogeneous colorectal lesions (>20 mm)
  Interventions: Procedure: Cold Snare Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Standard Endoscopic Mucosal Resection — Use of injected colloidal or saline solution to raise a lesion prior to polypectomy snare closed over a polyp with electrocautery
  Other Names: Standard EMR
  Arms: Standard Endoscopic Mucosal Resection
Procedure: Cold Snare Endoscopic Mucosal Resection — Use of injected colloidal or saline solution to raise a lesion prior to polypectomy snare closed over a polyp without electrocautery
  Other Names: Cold EMR
  Arms: Cold Snare Endoscopic Mucosal Resection

SUMMARY:
This study compares the effectiveness in complete resection (absence of recurrence at 6 months) the two different techniques for performing endoscopic mucosal resection (EMR) of nonpedunculated homogeneous colorectal lesions >20mm

DETAILED DESCRIPTION:
Colonoscopy is the reference diagnostic test for the study of colon diseases. This procedure also allows the realization of endoscopic therapeutics techniques; thus, endoscopic mucosal resection (EMR) is an effective and safe therapy for the treatment of premalignant and early malignant colorectal lesions of the colon and its use is universal.

Usually, colon lesions larger than 10 mm (or pedunculated of any size) require for resection the use of electrocoagulation current (or hot snare polypectomy) and thus is reflected in the most recent clinical practice guidelines (ESGE guidelines, for example). However, the risk of side adverse effects from the use of electrocoagulation is not insignificant and includes post-polypectomy bleeding, post-polypectomy syndrome, post-polypectomy fever and/or immediate or delayed perforation. This risk of complications is higher depending on the characteristics and size of colorectal lesions resected.

On the other hand, currently in small lesions not pedunculated (< 10 mm), it is recommended to use cold snare polypectomy according to ESGE clinical guidelines, as it has been seen in previous studies that this reduces complication rates without varying the effectiveness in resection.

However, in lesions > 10 mm the previous experience with cold snare resection is less, probably motivated by the possible drawbacks in terms of the possible difficulty of resection of thick tissue with cold snare and a possible increased intra-procedure hemorrhagic risk that can make it difficult to see the scar, with the possibility of leaving residual tissue.

However, in recent years the accumulated evidence gathered in various studies and grouped in a recent systematic review suggests that endoscopic mucosal resection with cold snare (Cold-EMR) may be safer than electrocoagulation resection for both 10-19mm lesions and for lesions >20 mm, associated with a lower rate of adverse effects with similar efficacy rates in terms of complete resection and adenomatous recurrence rate. Still, evidence for the treatment of nonpedunculated lesions >20 mm is relatively limited and is not based on randomized comparative studies with the standard EMR technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age > 18 years undergoing a colonoscopy for any reason of request and who do not meet exclusion criteria.
* Nonpedunculated homogeneous colorectal lesions type LST ( Paris 0-IIa morphology) and serrated lesions larger than 20 mm without endoscopic data of malignancy: NICE 1 pattern +/- NICE 2 component ( serrated lesions) or NICE2 pattern/JNET 2A (adenomas) and therefore subsidiaries of RME. Randomization will be performed per patient, not for colorectal lesions
* Signature of informed consent of endoscopic exploration

Exclusion Criteria:

* .No signature of informed consent prior to the study procedure.
* Absence of proper suspension of the anticoagulant/antiplatelet therapy prior to procedure according to usual pre-procedure recommendations (BSG and ESGE guidelines)
* Patients with severe thrombopenia/ coagulopathy (Platelets < 50,000/INR > 1.5) not corrected prior to procedure (plasma or platelet transfusion)
* Patients not candidates for endoscopic resection of colorectal lesions by comorbidities.
* Pregnant.
* Patients with inflammatory bowel disease (IBD)
* Urgent colonoscopy.
* Poor preparation (BBPS <2 in the colon segment where the lesion is located)
* Laterally spreading tumors (LST) lesions with non-homogeneous morphology including: sessile polyps (0-Is), pedunculated (0-Ip) and LST lesions with depressed or excavated components (Paris 0-IIc or Paris 0-III), LST granular nodular mixed, LST-G with whole nodular type. In case of doubt depressed component (Paris 0-IIc) or histological borderline lesion (JNET2B), will be excluded from the study.
* Histological prediction of deep invasive or non-subsidiary to endoscopic mucosal resection lesion as a treatment of choice: NICE 3 pattern by inspection with NBI or Kudo V pattern in traditional/electronic chromoendoscopy or Sano IIIA/IIIB pattern
* Endoscopic resection of post-EMR scar level relapses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Complete resection of the lesion | 3-6 months
  Complete resection of the lesion is defined as the non-visualization by the endoscopist of a residual lesion in the mucosal defect and its edge at the end of the EMR and no visualization of recurrence in the post-EMR scar on the first surveillance colonoscopy and absence of recurrence data in scar biopsies

SECONDARY OUTCOMES:
Security profile | 30 days
  Security profile is defined as the observed percentage of complications (Intra-procedure bleeding, deferred bleeding, deferred bleeding in antiplatelet and/or anticoagulated patients,post-polypectomy fever, post-polypectomy syndrome, deep muscle damage and perforation) in each of the evaluated techniques.
Late adenoma recurrence rate | 18 months
  Late adenoma recurrence rate as determined by endoscopic assessment (no visible recurrent adenoma) and histological assessment (scar biopsies) in surveillance colonoscopy at 18 months of the procedure
Number of fragments needed to complete the resection | 1 day
  Number of fragments needed to resect with polypectomy snare to complete the resection of the colorectal lesion.
Resection time | 1 day
  Time needed to perform endoscopic mucosal resection measured from first snare positioning until complete resection is achieved based on endoscopic assessment.
Bloc resection rate | 1
  Number of lesions that have undergone resection in a single fragment with each of these evaluated techniques.
R0 resection rate | 1 day
  Number of lesions with complete macroscopic resection with a negative microscopic margin in the mucosectomy specimen
EMR technique conversion rate | 1 day
  Number of lesions to be finally resected with the other arm of study technique not initially assigned
Need for additional treatments to complete the resection. | 1 day
  Number of lesions that cannot be completely resected with the assigned EMR technique, requiring different techniques to complete the resection, such as SOFT coagulation with snare tip, APC (argon plasma coagulation), hot avulsion with hot biopsy forceps, biopsy forceps, biopsy forceps +ablation
Number of clips used | 1 day
  Number of clip used for hemostatic purposes or for the prophylactic closure of the injury
Degree of artifact/interference in the histological interpretation | 1 day
  Subjective impression of the artifact in the histological interpretation of the resected sample (null, moderate, severe)
Depth of the resected submucosa | 1 day
  Measure the depth of the resected submucosa layer (in microns) with each of the resection techniques used
Percentage of mucosal muscle present in the mucosal protrusions in the resection defect of cold-EMR. | 1 day
  Assess the percentage of presence of mucosal muscle in biopsies performed on the protrusions present in the resection defect of cold-EMR
Need for surgery for technical failure | 6 months
  Number of lesions that have to be finally resected by surgery due to technical impossibility for their endoscopic resection.
Cost-effectiveness study. | 18 months
  evaluate the cost-effectiveness of each of the endoscopic mucosal resection techniques
Sub-analysis by center participating in the study | 18 months
  A subanalysis of the study results by center will be carried out to rule out significant differences between them

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Nogales, Principal Investigator — Hospital General Universitario Gregorio Marañon
Locations (1):
- Óscar Nogales Rincón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thoguluva Chandrasekar V, Spadaccini M, Aziz M, Maselli R, Hassan S, Fuccio L, Duvvuri A, Frazzoni L, Desai M, Fugazza A, Jegadeesan R, Colombo M, Dasari CS, Hassan C, Sharma P, Repici A. Cold snare endoscopic resection of nonpedunculated colorectal polyps larger than 10 mm: a systematic review and pooled-analysis. Gastrointest Endosc. 2019 May;89(5):929-936.e3. doi: 10.1016/j.gie.2018.12.022. Epub 2019 Jan 9. PMID 30639542
- [Background] Horiuchi A, Nakayama Y, Kajiyama M, Tanaka N, Sano K, Graham DY. Removal of small colorectal polyps in anticoagulated patients: a prospective randomized comparison of cold snare and conventional polypectomy. Gastrointest Endosc. 2014 Mar;79(3):417-23. doi: 10.1016/j.gie.2013.08.040. Epub 2013 Oct 11. PMID 24125514
- [Background] Takeuchi Y, Yamashina T, Matsuura N, Ito T, Fujii M, Nagai K, Matsui F, Akasaka T, Hanaoka N, Higashino K, Iishi H, Ishihara R, Thorlacius H, Uedo N. Feasibility of cold snare polypectomy in Japan: A pilot study. World J Gastrointest Endosc. 2015 Nov 25;7(17):1250-6. doi: 10.4253/wjge.v7.i17.1250. PMID 26634041
- [Background] Aslan F, Camci M, Alper E, Akpinar Z, Arabul M, Celik M, Unsal B. Cold snare polypectomy versus hot snare polypectomy in endoscopic treatment of small polyps. Turk J Gastroenterol. 2014 Jun;25(3):279-83. doi: 10.5152/tjg.2014.5085. PMID 25141316
- [Background] Tate DJ, Awadie H, Bahin FF, Desomer L, Lee R, Heitman SJ, Goodrick K, Bourke MJ. Wide-field piecemeal cold snare polypectomy of large sessile serrated polyps without a submucosal injection is safe. Endoscopy. 2018 Mar;50(3):248-252. doi: 10.1055/s-0043-121219. Epub 2017 Nov 23. PMID 29169195
- [Background] Hirose R, Yoshida N, Murakami T, Ogiso K, Inada Y, Dohi O, Okayama T, Kamada K, Uchiyama K, Handa O, Ishikawa T, Konishi H, Naito Y, Fujita Y, Kishimoto M, Yanagisawa A, Itoh Y. Histopathological analysis of cold snare polypectomy and its indication for colorectal polyps 10-14 mm in diameter. Dig Endosc. 2017 Jul;29(5):594-601. doi: 10.1111/den.12825. Epub 2017 May 17. PMID 28160332
- [Background] Rameshshanker R, Tsiamoulos Z, Latchford A, Moorghen M, Saunders BP. Resection of large sessile serrated polyps by cold piecemeal endoscopic mucosal resection: Serrated COld Piecemeal Endoscopic mucosal resection (SCOPE). Endoscopy. 2018 Jul;50(7):E165-E167. doi: 10.1055/a-0599-0346. Epub 2018 May 9. No abstract available. PMID 29742770
- [Background] Rex KD, Vemulapalli KC, Rex DK. Recurrence rates after EMR of large sessile serrated polyps. Gastrointest Endosc. 2015 Sep;82(3):538-41. doi: 10.1016/j.gie.2015.01.025. Epub 2015 Apr 4. PMID 25851161
- [Background] Qu J, Jian H, Li L, Zhang Y, Feng B, Li Z, Zuo X. Effectiveness and safety of cold versus hot snare polypectomy: A meta-analysis. J Gastroenterol Hepatol. 2019 Jan;34(1):49-58. doi: 10.1111/jgh.14464. Epub 2018 Sep 26. PMID 30176072
- [Background] Veitch AM, Vanbiervliet G, Gershlick AH, Boustiere C, Baglin TP, Smith LA, Radaelli F, Knight E, Gralnek IM, Hassan C, Dumonceau JM. Endoscopy in patients on antiplatelet or anticoagulant therapy, including direct oral anticoagulants: British Society of Gastroenterology (BSG) and European Society of Gastrointestinal Endoscopy (ESGE) guidelines. Endoscopy. 2016 Apr;48(4):c1. doi: 10.1055/s-0042-122686. Epub 2017 Jan 23. No abstract available. PMID 28114689
- [Background] Burgess NG, Bassan MS, McLeod D, Williams SJ, Byth K, Bourke MJ. Deep mural injury and perforation after colonic endoscopic mucosal resection: a new classification and analysis of risk factors. Gut. 2017 Oct;66(10):1779-1789. doi: 10.1136/gutjnl-2015-309848. Epub 2016 Jul 27. PMID 27464708
- [Background] Takayanagi D, Nemoto D, Isohata N, Endo S, Aizawa M, Utano K, Kumamoto K, Hojo H, Lefor AK, Togashi K. Histological Comparison of Cold versus Hot Snare Resections of the Colorectal Mucosa. Dis Colon Rectum. 2018 Aug;61(8):964-970. doi: 10.1097/DCR.0000000000001109. PMID 29944582
- [Background] Rodriguez Sanchez J, Sanchez Alonso M, Pellise Urquiza M. The "bubble sign": a novel way to detect a perforation after cold snare polypectomy. Endoscopy. 2019 Aug;51(8):796-797. doi: 10.1055/a-0881-2856. Epub 2019 May 9. No abstract available. PMID 31071753
- [Background] Keklikkiran C, Ozdogan OC. Thermal ablation of mucosal defect margins reduces adenoma recurrence after colonic endoscopic mucosal resection. Turk J Gastroenterol. 2019 Jun;30(6):580-581. doi: 10.5152/tjg.2019.210519. No abstract available. PMID 31144663
- [Background] Moss A, Williams SJ, Hourigan LF, Brown G, Tam W, Singh R, Zanati S, Burgess NG, Sonson R, Byth K, Bourke MJ. Long-term adenoma recurrence following wide-field endoscopic mucosal resection (WF-EMR) for advanced colonic mucosal neoplasia is infrequent: results and risk factors in 1000 cases from the Australian Colonic EMR (ACE) study. Gut. 2015 Jan;64(1):57-65. doi: 10.1136/gutjnl-2013-305516. Epub 2014 Jul 1. PMID 24986245
- [Derived] Nogales O, Carbonell Blanco C, Montori Pina S, Pellise M, Martinez Sempere JF, Riu Pons F, Mangas-Sanjuan C, Daca-Alvarez M, Uchima H, Aranda-Hernandez J, Alvarez Delgado A, Rodriguez de Santiago E, Santiago Garcia J, Canete Ruiz A, Miranda Garcia P, Nunez Rodriguez H, Herreros-de-Tejada A, Valdivielso Cortazar E, De Maria P, Busquets D, Elosua A, Rivero-Sanchez L, Lopez-Ibanez M, Alvarez-Gonzalez MA, Albeniz E; Mucosal Resection and Third-Space Endoscopy SEED Working Group. Cold snare endoscopic mucosal resection versus standard hot technique for large flat nonpedunculated colonic lesions: a randomized controlled trial. Endoscopy. 2025 Aug;57(8):851-861. doi: 10.1055/a-2542-9759. Epub 2025 Feb 19. PMID 39970943